CLINICAL TRIAL: NCT06971406
Title: A Multicenter, Prospective Phase II Clinical Study of High-Dose Firmonertinib Combined With Bevacizumab and Intrathecal Pemetrexed in the Treatment of EGFR-Mutated Non-Small Cell Lung Cancer With Leptomeningeal Metastasis
Brief Title: High-Dose Firmonertinib Combined With Bevacizumab and Intrathecal Pemetrexed in the Treatment of EGFR-Mutated Non-Small Cell Lung Cancer With Leptomeningeal Metastasis
Acronym: FLAME-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qiming Wang (Other Government)
Responsible Party: Sponsor-Investigator, Qiming Wang, professor and chair, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-083
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer; EGFR Mutation; Leptomeningeal Metastases; Targeted Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prospective cohort (Experimental): high-dose firmonertinib (240 mg, daily), bevacizumab (15 mg/kg, every 3 weeks), and pemetrexed (50 mg, intrathecal chemotherapy,C1 d1d5,then every 3 weeks)
  Interventions: Drug: Combination therapy prospective cohort

INTERVENTIONS:
Drug: Combination therapy prospective cohort — high-dose firmonertinib (240 mg, daily), bevacizumab (15 mg/kg, every 3 weeks), and pemetrexed (50 mg, intrathecal chemotherapy C1d1d5, then every 3 weeks)

SUMMARY:
Primary Objective:

To evaluate the efficacy of high-dose firmonertinib combined with bevacizumab and intrathecal pemetrexed in EGFR Ex19del/L858R-mutated non-small cell lung cancer (NSCLC) with leptomeningeal metastasis (LM), as measured by Overall Survival (OS).

Secondary Objectives:

1. To assess the efficacy of this regimen in EGFR Ex20ins/PACC/L861Q-mutated NSCLC with LM.
2. To further evaluate therapeutic outcomes across cohorts, including:

   * Time to Treatment Failure (TTF)
   * Leptomeningeal Objective Response Rate (ORR-LM)
   * Clinical Response Rate
3. To analyze the impact of this regimen on *quality of life* using standardized metrics:

   * EORTC QLQ-C30
   * EORTC QLQ-LC13
4. To assess safety profiles across cohorts, focusing on:

   * Incidence and severity of adverse events (AEs) graded per *CTCAE v5.0*
   * Frequency of treatment-related toxicities

Exploratory Objectives:

To investigate correlations between dynamic changes in:

* Plasma-derived circulating tumor DNA (ctDNA)
* Cerebrospinal fluid-derived cell-free DNA (cfDNA) and clinical outcomes through comparative analysis of genomic profiling and epigenetic signatures before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have obtained written informed consent from the patient or his or her legal representative.
2. Age ≥18 years, male or female.
3. Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC).
4. EGFR mutations confirmed by genetic testing (EGFR Ex19del/L858R/Ex20ins/PACC/L861Q).
5. Leptomeningeal metastasis diagnosed by comprehensive clinical assessment according to "EANO-ESMO" diagnostic criteria, including symptom evaluation, imaging assessment, and/or cerebrospinal fluid (CSF) cytopathological evaluation.
6. Both treatment-naïve leptomeningeal metastasis patients and those who progressed after standard antitumor therapies in clinical practice are eligible. ≤3 prior lines of therapy allowed (patients with >3 prior lines may enroll in the real-world study cohort).
7. ECOG PS 0-2 (patients with ECOG PS >2 may enroll in the real-world study cohort).
8. Prior radiotherapy or surgical treatment targeting the central nervous system (CNS) is permitted.
9. Patients with CNS symptoms/signs are allowed if these manifestations are not life-threatening.
10. Patients previously treated with standard-dose third-generation EGFR TKIs, pemetrexed intravenous infusion, or bevacizumab are permitted.
11. Adequate organ function:

    Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥80g/L Total bilirubin ≤1.5×ULN, AST/ALT ≤2.5×ULN (≤3×ULN for bilirubin and ≤5×ULN for AST/ALT in cases with liver metastasis) Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula).
12. Sexually active males or females of childbearing potential must use highly effective contraception (e.g., oral contraceptives, IUD, abstinence, or barrier methods with spermicide) during the trial and for 12 months after treatment completion.

Exclusion Criteria:

1. Diagnosis of other malignancies within the past 5 years or history of other malignancies (except adequately controlled basal cell carcinoma of the skin, cervical carcinoma in situ, or ductal carcinoma in situ of the breast).
2. Severe gastrointestinal disorders affecting drug administration or absorption, including but not limited to peptic ulcer disease, inflammatory bowel disease, etc.
3. Known or suspected hypersensitivity to the investigational drugs (Firmonertinib, Bevacizumab, Pemetrexed) or any of their excipients.
4. Prior treatment with high-dose third-generation EGFR TKI or intrathecal chemotherapy with Pemetrexed.
5. Evidence of any severe or uncontrolled systemic diseases, including uncontrolled hypertension, diabetes, active bleeding, or active infections (e.g., hepatitis B/C, HIV), which in the investigator's judgment may jeopardize patient participation or protocol compliance.
6. History of steroid-requiring radiation pneumonitis or any evidence of active interstitial lung disease.
7. Clinically significant cardiac arrhythmias (e.g., QTc interval >500 ms) or heart failure (left ventricular ejection fraction <50%).
8. Pregnant or lactating women.
9. Patients currently participating in or having received investigational drug therapy within 2 weeks prior to enrollment.
10. Other severe acute/chronic medical or psychiatric conditions or laboratory abnormalities that, in the investigator's opinion, may increase study-related risks, interfere with result interpretation, or compromise the patient's ability to complete the study or adhere to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
OS（EGFR Ex19del/L858R） | the time between the date of enrollment and the date of death from any cause for EGFR Ex19del/L858R NSCLC with leptomeningeal metastases(up to 36 months)
  overall survive time （EGFR Ex19del/L858R）

SECONDARY OUTCOMES:
OS（EGFREx20ins/PACC/L861Q） | the time between the date of enrollment and the date of death from any cause for EGFREx20ins/PACC/L861Q NSCLC with leptomeningeal metastases(up to 36 months)
  overall survive time（EGFREx20ins/PACC/L861Q）
TTF | up to 24 months
  time to treatment failure:The time interval from the start of the triple therapy to treatment failure
ORR-LM | up to 24 months
  Objective Response Rate in Leptomeningeal Metastases：the proportion of patients whose leptomeningeal lesions achieve a complete response (CR) or partial response (PR) during the study period from the first administration of the study drug until leptomeningeal disease progression
CRR | up to 24 months
  Clinical response rate：the proportion of patients whose CR, OR, or PR lasts for at least one week
Quality of life assessment (EORTC QLQ-C30, EORTC QLQ-LC13) | At the end of every 2 cycles(each cycle is 21 days)
  EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire - 30 items, score:30-126, Higher scores indicate worse quality of life) and EORTC QLQ-LC13(European Organization for Research and Treatment of Cancer Quality of Life Lung Module 13 items) were used to assess the quality of life, scores were normalized to 0-100, with high scores in the symptom domain indicating severe symptoms and high scores in the functional domain indicating good functioning
AE | At the end of every 2 cycles(each cycle is 21 days)
  AEs (Adverse events)were graded according to CTCAE v5.0 every two cycles after enrollment

IPD SHARING:
Plan to Share IPD: No